CLINICAL TRIAL: NCT02557321
Title: A Phase 1b/2 Study of PV-10 Intralesional Injection in Combination With Systemic Immune Checkpoint Inhibition for Treatment of Metastatic Melanoma
Brief Title: PV-10 in Combination With Pembrolizumab for Treatment of Metastatic Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Provectus Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Provectus Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-MM-1201
Record Dates: First submitted 2015-09-20; First posted 2015-09-23 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Rose Bengal B; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1b (Experimental): PV-10 (intralesional) and pembrolizumab (2 mg/kg every 3 weeks)
  Interventions: Drug: PV-10; Drug: Pembrolizumab
- Phase 2 (Arm 1) (Experimental): PV-10 (intralesional) and pembrolizumab (2 mg/kg every 3 weeks)
  Interventions: Drug: PV-10; Drug: Pembrolizumab
- Phase 2 (Arm 2) (Active Comparator): Pembrolizumab (2 mg/kg every 3 weeks)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: PV-10 — PV-10 will be administered by intralesional injection every 3 weeks at Day 1 (Week 1), Week 4, Week 7, Week 10 and Week 13
  Other Names: Rose Bengal Disodium
  Arms: Phase 1b; Phase 2 (Arm 1)
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously every 3 weeks starting at Day 1 (Week 1)

SUMMARY:
This is an international multicenter, open-label, sequential phase study of intralesional (IL) PV-10 in combination with immune checkpoint inhibition. Metastatic melanoma patients (Stage IV or Stage III unresectable, in-transit or satellite disease) with at least one injectable lesion who are candidates for pembrolizumab (both treatment naïve patients and treatment refractory patients who have failed to achieve a complete or partial response to or previously progressed on one or more checkpoint inhibitor) will be eligible for study participation. In the Phase 1b portion of the study, all participants will receive the combination of IL PV-10 and pembrolizumab (i.e., PV-10 + standard of care). In the subsequent Phase 2 portion of the study participants will be randomized 1:1 to receive either the combination of IL PV-10 and pembrolizumab or pembrolizumab alone (i.e., PV-10 + standard of care vs. standard of care).

DETAILED DESCRIPTION:
Phase 1b. Up to 24 eligible subjects will be enrolled in an initial cohort in the Phase 1b portion of the study (Main Cohort). Up to an additional 24 eligible subjects who have failed to achieve a complete or partial response to or progressed on prior checkpoint inhibition will be enrolled in a first expansion cohort (Expansion Cohort 1). Up to an additional 24 eligible subjects with Stage III unresectable, in-transit or satellite melanoma will be enrolled in a second expansion cohort (Expansion Cohort 2). Each subject in each Phase 1b cohort will receive the combination of IL PV-10 and pembrolizumab.

Phase 2. A total of an estimated 120 eligible subjects will be randomized in a 1:1 ratio to the two treatment arms (i.e., PV-10 + pembrolizumab or pembrolizumab alone) in the Phase 2 portion of the study. This number of subjects may be modified based on emerging evidence of preliminary efficacy and effect size from the Phase 1b and initial Phase 2 portions of the study.

Subjects assigned to receive PV-10 in Phase 1b and 2 will receive initial IL PV-10 to their injectable lesions commencing on study Day 1 for up to 12 weeks (i.e., investigational Treatment Phase of the study). PV-10 may be re-administered at 21-day (3-week) intervals during the Treatment Phase of the study to any remaining, uninjected injectable lesions until all injectable lesions have been injected. Lesions that fail to exhibit complete ablation may be re-injected on this schedule.

Pembrolizumab will be administered at 21-day (3-week) intervals per prescribing information (label) commencing on study Day 1 for up to 24 months or until disease progression, toxicity requiring discontinuation of study treatment or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, male or female.
2. Histologically or cytologically confirmed diagnosis of melanoma.
3. Stage IV or Stage III (unresectable, in-transit or satellite) melanoma.
4. At least 1 Injectable Lesion (i.e., cutaneous, subcutaneous, soft tissue, superficial nodal or palpable nodal lesion with longest diameter at least 5 mm that is suitable for injection with PV-10).
5. A minimum of 1 measurable Target Lesion that can be accurately measured by calipers, computed tomography (CT) or magnetic resonance imaging (MRI) consisting of at least one of the following:

   * at least one cutaneous lesion (each lesion ≥ 10 mm longest diameteror up to 5 lesions in aggregate having a sum of longest diameters ≥ 10 mm); and/or
   * at least one subcutaneous or soft tissue lesion (each lesion ≥ 10 mm in longest diameter by CT or MRI); and/or
   * at least one nodal lesion (each lesion ≥ 15 mm in short axis diameter by CT or MRI); and/or
   * at least one visceral lesion (each lesion ≥ 10 mm in longest diameter by CT or MRI).
6. Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1.
7. Clinical Laboratories:

   * absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥100 x 109/L
   * estimated creatinine clearance (CrCl, by Cockcroft-Gault formula) or estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2
   * total bilirubin ≤ 3 times the upper limit of normal (ULN)
   * aspartate transaminase (AST), alanine transaminase (ALT) and alkaline phosphatase (ALP) ≤ 5 times the upper limit of normal (ULN)
8. Thyroid function abnormality ≤ Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2.

Exclusion Criteria:

1. Untreated or clinically active melanoma brain metastases.

   * Subjects with ≤ 3 brain metastases and each ≤ 1 cm size that were treated with either surgical resection and/or radiation therapy are eligible for study participation provided (a) there is no evidence of progressive central nervous system (CNS) disease on brain imaging at least 30 days after definitive treatment and (b) the subject is not taking prednisone at >10 mg or equivalent daily.
   * Subjects with > 1 cm or > 3 in number treated brain metastases are eligible for study participation provided (a) there is no evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy and (b) if the subject is not taking prednisone at >10 mg or equivalent daily.
2. Prior treatment with PV-10 or any checkpoint inhibitor; however, subjects (a) who have failed to achieve a complete or partial response within 24 weeks following initiation of checkpoint inhibition or (b) who progressed after more than 12 weeks of checkpoint inhibition are eligible for study participation in the Phase 1b Expansion Cohort 1 without washout period for checkpoint inhibition.
3. Other prior cancer therapy or anti-cancer vaccine within the lesser of 4 weeks or 5 half-lives before initial study treatment.
4. Known sensitivity to any of the products or components to be administered during dosing.
5. Concurrent or Intercurrent Illness:

   * History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other systemic autoimmune disease.
   * Evidence of clinically significant immunosuppression.
   * Impaired wound healing or other extremity complications due to severe or uncontrolled diabetes mellitus in subjects whose Injectable Lesions are located in an extremity.
   * Severe peripheral vascular disease (i.e., severe claudication [pain occurring after less than 200 meters of walking], rest pain, ischemic ulceration or gangrene) in subjects whose Injectable Lesions are located in an extremity.
   * Significant concurrent or intercurrent illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the Investigator, compromise the subject's safety or compliance or interfere with interpretation of study results.
   * Uncontrolled thyroid disease or cystic fibrosis.
   * Clinically significant acute or unstable cardiovascular, cerebrovascular (stroke), renal, gastrointestinal, pulmonary, immunological, endocrine, or central nervous system disorders.
   * Malignancy other than melanoma within 2 years of enrollment except for: adequately treated (i.e., with curative intent) basal or squamous cell carcinoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer.
6. Pregnancy:

   * Female subjects who are pregnant or lactating.
   * Female subjects who have positive serum pregnancy test taken within 14 days of initiation of study treatment.
   * Female subjects of childbearing potential (defined as having a menstrual cycle within the past 12 months and not having had a surgical procedure to accomplish sterilization) who are not using highly effective contraception (e.g., oral contraceptives, intrauterine devices, double barrier methods such as condoms and diaphragms, abstinence or equivalent measures).
   * Male subjects who are unwilling to use acceptable method of effective contraception.
7. Subjects unable to comprehend and give informed consent are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the combination regimen assessed by adverse events (AEs) | Start of treatment until 4 weeks after final administration of PV-10
  Phase 1b: Safety and tolerability of the combination regimen will be assessed by monitoring the frequency, duration, severity and attribution of adverse events (AEs) and toxicities requiring discontinuation of study treatment, and evaluating changes in laboratory values and vital signs
Progression Free Survival (PFS) | Up to 24 months from initiation of study treatment
  Phase 2: Response evaluated by blinded independent review committee assessment per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months from initiation of study treatment
  Phase 1b: Response evaluated per RECIST 1.1
Objective Response Rate (ORR) | Up to 24 months from initiation of study treatment
  Phase 1b and 2: Response evaluated per RECIST 1.1
Change in immune biomarkers | Up to 28 weeks from initiation of study treatment
  Phase 1b: Peripheral Blood Mononuclear Cells (PBMCs) assessed vs. baseline values for changes in T cell populations
Overall Survival (OS) | 24 months from initiation of study treatment for last subject randomized
  Phase 1b and 2
Safety and tolerability of the combination regimen assessed by adverse events (AEs) | Start of treatment until 4 weeks after final administration of PV-10
  Phase 2: Safety and tolerability of the combination regimen will be assessed by monitoring the frequency, duration, severity and attribution of adverse events (AEs) and toxicities requiring discontinuation of study treatment, and evaluating changes in laboratory values and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health & Science University, Portland, Oregon
  - St Luke's University Health Network, Easton, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas